CLINICAL TRIAL: NCT07163637
Title: A Randomized, Double-Blind, Placebo-Controlled Decentralized Trial to Assess the Effect and Tolerability of Limosilactobacillus Reuteri DSM 17648 Supplement in Healthy Adults Reporting Upper Gastrointestinal Discomfort
Brief Title: Effect of Limosilactobacillus Reuteri DSM 17648 in Healthy Adults Reporting Upper Gastrointestinal Discomfort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HHB-IM-24-07
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants; Upper Gastrointestinal Discomfort

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limosilactobacillus reuteri DSM 17648 (Experimental): Participant will take one capsule of L. reuteri DSM 17648 once per day with liquid during or immediately after the main meal, for 8 weeks.
  Interventions: Dietary Supplement: Limosilactobacillus reuteri DSM 17648
- Placebo (Placebo Comparator): Participant will take one capsule of placebo once per day with liquid during or immediately after the main meal, for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Limosilactobacillus reuteri DSM 17648 — One capsule containing L. reuteri DSM 17648 should be taken once per day with liquid during or immediately after the main meal, for 8 weeks.
  Other Names: Pylopass; PyloGuard
  Arms: Limosilactobacillus reuteri DSM 17648
Dietary Supplement: Placebo — One capsule of placebo should be taken once per day with liquid during or immediately after the main meal, for 8 weeks.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the food supplement containing a postbiotic (inanimate) Limosilactobacillus reuteri DSM 17648 works to improve the symptoms of upper gastrointestinal discomfort in healthy adults. The main questions it aims to answer are:

1. Does L. reuteri DSM 17648 reduce the frequency of the symptoms of upper gastrointestinal discomfort, including acid reflux-related and dyspeptic symptoms, and its relief rate, over 8 weeks of intake?
2. Does L. reuteri DSM 17648 improve gastrointestinal-related quality of life, and perceived stress?
3. How well do participants tolerate the L. reuteri DSM 17648 supplement?
4. Does L. reuteri DSM 17648 have an effect on the gut microbiota? (Exploratory aim)

Researchers will compare supplement containing L. reuteri DSM 17648 to a placebo (a look-alike supplement capsule that contains no L. reuteri DSM 17648).

Participants will:

* Take L. reuteri DSM 17648 supplement or a placebo every day for 8 weeks
* Answer questionnaires once every 2 weeks
* Provide stool samples for microbiome assessment at 2 timepoints (baseline and end of study (8 weeks))
* provide weekly information on investigational product intake and any adverse event records

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female.
2. Anyone with a BMI less than or equal to 32 kg/m².
3. Be aged 30-70.
4. Anyone currently experiencing occasional upper gastrointestinal discomfort (approximately 2 times/week over the past month), including the following:

   1. Heartburn
   2. Upper abdominal pain
   3. Reflux
   4. Pain or burning in the stomach
5. Anyone with an FSSG (Frequency Scale for the Symptoms of GERD) total score of 8 or above.
6. Anyone who is generally healthy - does not live with any uncontrolled chronic health conditions, such as cancer, mental health disorders, history of serious illness in the last three months, history of substance abuse, or planned surgery during the study period.
7. Willing to avoid introducing any new supplements, over-the-counter medications, or herbal remedies for the duration of this trial
8. If taking other supplements, over-the-counter medications, or herbal remedies unrelated to gut health, has been doing so consistently for a minimum of three months.
9. Willing to maintain current diet, sleep pattern, and activity levels for the duration of the trial.
10. Resides in the United States.

Exclusion Criteria:

* 1. Anyone with any allergies or sensitivities to any of the study product ingredients.

  2. Any women who are pregnant, breastfeeding, or trying to conceive (or who will be at any point during the study period).

  3. Anyone unwilling to follow the study protocol. 4. Anyone taking any supplement, over-the-counter medication, or herbal remedy targeting gut health.

  5. Anyone with a known history of severe digestive disorders like GERD (Gastroesophageal Reflux Disease) and FD (Functional Dyspepsia), Irritable Bowel Syndrome (IBS), Irritable Bowel Disease (IBD), Crohn's disease, celiac disease, chronic constipation, chronic diarrhea, or gastrointestinal tract disorders or surgeries.

  6. Anyone currently or recently (within the past 2 weeks) taking probiotic foods, including yoghurts.

  7. Anyone currently or recently (within the last 12 weeks) taking medication, including proton pump inhibitors, anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, monoamine oxidase inhibitors (MAOIs), or thyroid products.

  8. Currently partaking in another research study or will partake in any other research study for the next eight weeks or at any point during this study's duration.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the total score of Frequency Scale for the Symptoms of GERD (FSSG) at 8 weeks | Baseline; 8 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG questionnaire comprises twelve questions in two domains, i.e. the acid reflux related symptom domain and dyspeptic symptom domain. The FSSG uses a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. Total FSSG score ranges from 0-48. Higher score indicates higher frequency.

SECONDARY OUTCOMES:
Change from Baseline in the total score of Frequency Scale for the Symptoms of GERD (FSSG) at 2 weeks | Baseline, 2 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG questionnaire comprises twelve questions in two domains, i.e. the acid reflux related symptom domain and dyspeptic symptom domain. The FSSG uses a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. Total FSSG score ranges from 0-48. Higher score indicates higher frequency.
Change from Baseline in the total score of Frequency Scale for the Symptoms of GERD (FSSG) at 4 weeks | Baseline, 4 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG questionnaire comprises twelve questions in two domains, i.e. the acid reflux related symptom domain and dyspeptic symptom domain. The FSSG uses a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. Total FSSG score ranges from 0-48. Higher score indicates higher frequency.
Change from Baseline in the total score of Frequency Scale for the Symptoms of GERD (FSSG) at 6 weeks | Baseline, 6 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG questionnaire comprises twelve questions in two domains, i.e. the acid reflux related symptom domain and dyspeptic symptom domain. The FSSG uses a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. Total FSSG score ranges from 0-48. Higher score indicates higher frequency.
Change from Baseline in the acid reflux related symptom sub-score of Frequency Scale for the Symptoms of GERD (FSSG) at 2 weeks | Baseline, 2 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG acid reflux related symptom sub-score domain comprises 7 questions, with answers in a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. FSSG acid reflux related symptom score ranges from 0-28. Higher score indicates higher frequency.
Change from Baseline in the acid reflux related symptom sub-score of Frequency Scale for the Symptoms of GERD (FSSG) at 4 weeks | Baseline, 4 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG acid reflux related symptom sub-score domain comprises 7 questions, with answers in a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. FSSG acid reflux related symptom score ranges from 0-28. Higher score indicates higher frequency.
Change from Baseline in the acid reflux related symptom sub-score of Frequency Scale for the Symptoms of GERD (FSSG) at 6 weeks | Baseline, 6 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG acid reflux related symptom sub-score domain comprises 7 questions, with answers in a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. FSSG acid reflux related symptom score ranges from 0-28. Higher score indicates higher frequency.
Change from Baseline in the acid reflux related symptom sub-score of Frequency Scale for the Symptoms of GERD (FSSG) at 8 weeks | Baseline, 8 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG acid reflux related symptom sub-score domain comprises 7 questions, with answers in a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. FSSG acid reflux related symptom score ranges from 0-28. Higher score indicates higher frequency.
Change from Baseline in the dyspeptic symptom sub-score of Frequency Scale for the Symptoms of GERD (FSSG) at 2 weeks | Baseline, 2 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG dyspeptic symptom sub-score domain comprises 5 questions, with answers in a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. FSSG dyspeptic symptom score ranges from 0-20. Higher score indicates higher frequency.
Change from Baseline in the dyspeptic symptom sub-score of Frequency Scale for the Symptoms of GERD (FSSG) at 4 weeks | Baseline, 4 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG dyspeptic symptom sub-score domain comprises 5 questions, with answers in a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. FSSG dyspeptic symptom score ranges from 0-20. Higher score indicates higher frequency.
Change from Baseline in the dyspeptic symptom sub-score of Frequency Scale for the Symptoms of GERD (FSSG) at 6 weeks | Baseline, 6 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG dyspeptic symptom sub-score domain comprises 5 questions, with answers in a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. FSSG dyspeptic symptom score ranges from 0-20. Higher score indicates higher frequency.
Change from Baseline in the dyspeptic symptom sub-score of Frequency Scale for the Symptoms of GERD (FSSG) at 8 weeks | Baseline, 8 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The FSSG dyspeptic symptom sub-score domain comprises 5 questions, with answers in a 5-point Likert scale (0-4) for each question, where: never = 0; occasionally = 1; sometimes = 2; often = 3; and always = 4. FSSG dyspeptic symptom score ranges from 0-20. Higher score indicates higher frequency.
Frequency Scale for the Symptoms of GERD (FSSG) relief rate at 4 weeks | Baseline, Week 4
  Relief rate is the number of participants whose symptoms were alleviated (lower score) at 4 weeks compared to Baseline based on the changes in FSSG scores.
Frequency Scale for the Symptoms of GERD (FSSG) relief rate at 8 weeks | Baseline, Week 8
  Relief rate is the number of participants whose symptoms were alleviated (lower score) at 8 weeks compared to Baseline based on the changes in FSSG scores.
Change from baseline quality of life, measured by Digestion-associated Quality of Life Questionnaire (DQLQ) at 2 weeks | Baseline, 2 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. DQLQ includes 9 statements that assess how often digestive events and experiences affected the quality of life over the past 7 days, with each scored on a 7-point Likert scale (Never = 0, Rarely = 0.1, Occasionally = 0.3, Sometimes = 0.5, Frequently = 0.7, Usually = 0.9, Always = 1.0). The total score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life.
Change from baseline quality of life, measured by Digestion-associated Quality of Life Questionnaire (DQLQ) at 4 weeks | Baseline, 4 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. DQLQ includes 9 statements that assess how often digestive events and experiences affected the quality of life over the past 7 days, with each scored on a 7-point Likert scale (Never = 0, Rarely = 0.1, Occasionally = 0.3, Sometimes = 0.5, Frequently = 0.7, Usually = 0.9, Always = 1.0). The total score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life.
Change from baseline quality of life, measured by Digestion-associated Quality of Life Questionnaire (DQLQ) at 6 weeks | Baseline, 6 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. DQLQ includes 9 statements that assess how often digestive events and experiences affected the quality of life over the past 7 days, with each scored on a 7-point Likert scale (Never = 0, Rarely = 0.1, Occasionally = 0.3, Sometimes = 0.5, Frequently = 0.7, Usually = 0.9, Always = 1.0). The total score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life.
Change from baseline quality of life, measured by Digestion-associated Quality of Life Questionnaire (DQLQ) at 8 weeks | Baseline, 8 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. DQLQ includes 9 statements that assess how often digestive events and experiences affected the quality of life over the past 7 days, with each scored on a 7-point Likert scale (Never = 0, Rarely = 0.1, Occasionally = 0.3, Sometimes = 0.5, Frequently = 0.7, Usually = 0.9, Always = 1.0). The total score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life.
Change from baseline perceived stress, measured by Perceived Stress Scale, at 4 weeks | Baseline, 4 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The 10-item Perceived Stress Scale (PSS-10) uses a 5-point Likert scale ranging from 0 (Never) to 4 (Very Often), with some items (positive worded items) reverse-scored to balance the scale. Total scores range from 0 to 40, with higher scores indicating higher levels of stress.
Change from baseline perceived stress, measured by Perceived Stress Scale, at 8 weeks | Baseline, 8 weeks
  Difference between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared. The 10-item Perceived Stress Scale (PSS-10) uses a 5-point Likert scale ranging from 0 (Never) to 4 (Very Often), with some items (positive worded items) reverse-scored to balance the scale. Total scores range from 0 to 40, with higher scores indicating higher levels of stress.
Number of participants with self-reported adverse events | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  Number of participants with self-reported adverse events will be collected and summarized descriptively at each time point for both the Limosilactobacillus reuteri DSM 17648 and placebo groups.

OTHER OUTCOMES:
Change from baseline microbiome profile in fecal samples at 8 weeks | Baseline, 8 weeks
  Difference in microbial diversity of fecal samples between Limosilactobacillus reuteri DSM 17648 and placebo arm will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Swathi Varanasi, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No